CLINICAL TRIAL: NCT03890458
Title: Effects of Vitamin D Supplements on Pregnancy Outcomes in Embriyo Transfer Cycles
Brief Title: The Effect of Vitamin D on Fertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Infertility; Infertility, Female; Vitamin D Deficiency; Vitamin D3 Deficiency
Keywords: vitamin D; vitamin D supplementation; infertility; D vitamin deficiency; infertile women; embryo transfer; pregnancy rate
MeSH Terms: conditions — Infertility; Infertility, Female; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: DEVIT-3
- Control (No Intervention)

INTERVENTIONS:
Drug: DEVIT-3 — The physicians gave the women in the experimental group vitamin D oral drops in an ampoule of 300,000 IU and a vial of 50,000 IU to take during the IVF treatment. Written and verbal information about how to take vitamin D was provided to the participants by the nurses. The women took 300,000 IU vitamin D orally for the first week. In the second week of the treatment, 50,000 IU vitamin D (15 drops/day) was used as maintenance dose until the pregnancy test day.
  Arms: Experimental

SUMMARY:
Objective: To examine the effect of vitamin D supplements on the pregnancy and clinical pregnancy rate in embryo transfer cycles.

Design: Experimental study with a pre- and post-test. Setting: In Vitro Fertilization Center Patients: Its sample consisted of 118 women, 58 in the experimental group and 60 in the control group.

Intervention(s): At the beginning of the infertility treatment, the experimental group took vitamin D supplements, and the control group did not. Vitamin D supplementation for infertile women includes regulation of a diet rich in vitamin D, educational and motivational interviews about insolation, and taking vitamin D orally.

Main Outcome Measure(s): 25(OH)D and beta HCG levels

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* literate in Turkish
* voluntary participation
* primarily infertile
* had undergone controlled ovarian hyperstimulation and had a fresh ET
* vitamin D levels lower than 30ng/mL before infertility treatment

Exclusion Criteria:

* patients with uncorrected congenital or acquired uterine anomalies
* bone, parathyroid gland, kidney and liver disorders
* use of anticonvulsants/antacid drugs
* taking dietary supplements contain vitamin D
* secondary infertility

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Blood Vitamin D level | The 25 (OH)D levels of the experimental group women were tested on the second or third day of their menstrual cycle. (Pretest)
  The vitamin D blood test was measured by the level of 25(OH)D.
Blood Vitamin D level | The 25 (OH)D levels of the women were tested on the two weeks after embryo transfer. (Posttest)
  The vitamin D blood test was measured by the level of 25(OH)D.

SECONDARY OUTCOMES:
Biochemical pregnancy | HCG levels of the women were evaluated on the two weeks after embryo transfer (Post test)
  The pregnancy test was measured level of HCG in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Teskereci, Principal Investigator — Akdeniz University
Locations (1):
- Murat Özekinci, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No